CLINICAL TRIAL: NCT03249727
Title: Analysis of Natural Killer Cell Activity (NKA) in Whole Blood in High Risk Subjects Undergoing Colonoscopy
Acronym: ANKA-HR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruiting issues
Sponsor: ATGen Canada Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: ANKA-HR
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Immunity, Innate; Colorectal Cancer
Keywords: natural killer cells; natural killer cell activity
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: All subjects will have a FIT (OC FIT-CHEK, Polymedco) and NK Vue test prior to colonoscopy
Who Masked: Outcomes Assessor
Masking Description: Endoscopist will not be provided the results of either the FIT or NK Vue tests performed as part of the trial; biochemist will not be provided the results of the colonoscopy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: IVDD for NK cell activity in whole blood — Once subject has been scheduled for a colonoscopy by the institution (up to 4 weeks prior to procedure), the subject will perform a FIT at home and an NK Vue test (one sample of one mL of blood) at the institution, prior to the day of colonoscopy.
  Other Names: NK Vue

SUMMARY:
This study will measure the activity of natural killer (NK) cells using the in vitro diagnostic device NK Vue in high risk subjects (Quebec risk categories P2, P3 and P4) scheduled for colonoscopy.

DETAILED DESCRIPTION:
In Quebec, subjects in risk category P2 are scheduled for colonoscopy due to high suspicion of cancer based on imaging, sigmoidoscopy or clinical exam. Subjects in categories P3 and P4 are scheduled for colonoscopy for one of the following reasons: suspicion of having an inflammatory bowel condition, rectal bleeding, presence of occult blood in stool, unexplained iron deficiency anemia, recent change in bowel habits, family history of CRC or adenomatous polyps or other hereditary colorectal diseases. Often, colonoscopy is not performed within the government-prescribed recommended delays, leading to waiting lists for the procedure. Analysis of NK cell activity may help identify those at risk for the presence of CRC and therefore help prioritize subjects on these waiting lists, help manage resources and help convince subjects to have a colonoscopy. Furthermore, all subjects will undergo a FIT, allowing a determination of the ability of each test alone, as well as a combination of NK Vue and FIT, to predict outcome on colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 40 and over who are scheduled to undergo colonoscopy at the research site and who are classified in category P2, P3 or P4.
2. Subjects who provide informed consent to participate in the trial

Exclusion Criteria:

1. Lack of understanding and/or participation due to illiteracy or inability to comprehend English or French
2. Subjects in category P3 who are there due to knowledge or suspicion of an inflammatory bowel disease
3. Previous history of cancer (any type) or active infection (as declared by the subject at the time of enrolment)
4. Currently participating (or participated within the previous 120 days) in an investigational therapeutic study (in case of interference of the drug with the immune system)
5. Subjects who underwent their colonoscopy and

   1. the colonoscopy preparation was judged insufficient
   2. the colonoscopy itself was judged insufficient or incomplete by the doctor
   3. the biopsy sample was lost and cancer could not be pathologically confirmed
   4. the colonoscopy detected an inflammatory bowel disease
6. Female who is pregnant, nursing, or of child-bearing potential while not practicing effective contraceptive methods.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
Test performance of NK Vue (ability of NK Vue to detect CRC in those subjects in risk categories P2, P3 or P4) | NK Vue blood draw taken within 7 days of FIT stool sampling and prior to colonoscopy
  Test performance of NK Vue for CRC will be assessed by ROC analysis and logistic regression, adjusting for subject baseline characteristics

SECONDARY OUTCOMES:
Test performance of FIT, to be determined at different cut-offs reflective of the various Canadian provincial cut-offs. | FIT performed at home and sample brought to institution within 7 days of collection and prior to coloscopy
  Test performance of FIT for CRC, using different cut-offs (≥50 ng/mL, ≥ 75 ng/mL, ≥ 100 ng/mL and ≥ 175 ng/mL), will be assessed by calculating the RR and by using ROC analyses at the different cut-offs.
Test performance of NK Vue in combination with FIT | FIT and NK Vue performed up to 4 weeks prior to colonoscopy, with NK Vue draw within 7 days of stool sampling
  Test performance of the combination of FIT at the different cut-offs (≥50 ng/mL, ≥ 75 ng/mL, ≥ 100 ng/mL and ≥ 175 ng/mL) and NK Vue (cut-off of <200 pg/mL), for CRC, will be assessed by calculating the RR and by using ROC analyses. Similar analyses will be done with subjects having either a positive FIT (at different cut-offs) or a NK Vue of <200 pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Jobin, MD, FRCP, Principal Investigator — CIUSSS de l'Est-de-l'île-de-Montréal; Installation Hôpital Maisonneuve-Rosemont
Locations (3):
- Canada (3):
  - CIUSSS de l'Est-de-l'île-de-Montréal, Installation Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - McGill University and the McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jobin G, Rodriguez-Suarez R, Betito K. Association Between Natural Killer Cell Activity and Colorectal Cancer in High-Risk Subjects Undergoing Colonoscopy. Gastroenterology. 2017 Oct;153(4):980-987. doi: 10.1053/j.gastro.2017.06.009. Epub 2017 Jun 15. PMID 28625834